CLINICAL TRIAL: NCT02339805
Title: Assessment of the Minimal Residual Disease in Diffuse Large B-Cell Lymphomas (DLBCL) From Cell-free Circulating DNA by Next Generation Sequencing (NGS)
Brief Title: Assessment of the Minimal Residual Disease in DLBCL From Cell-free Circulating DNA by NGS
Acronym: LymphoSeq
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Collaborators: U918 ( Inserm unit) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB13.03
Record Dates: First submitted 2015-01-13; First posted 2015-01-15 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Non Hodgkin Lymphoma
Keywords: Minimal residual disease, NGS, NHL, DNA sequencing
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasm, Residual | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- next generation sequencing (Experimental): Determination of clonotypic evolution of the minimal residual disease by next generation sequencing.
  Interventions: Other: next generation sequencing; Device: Fluorine-18 fluorodeoxyglucose positron emission tomography (18F-FDG-PET)

INTERVENTIONS:
Other: next generation sequencing — DNA from plasma, peripheral blood mononuclear cell and bone marrow will be sequenced by NGS for a panel of 34 genes.
Device: Fluorine-18 fluorodeoxyglucose positron emission tomography (18F-FDG-PET) — tumor Assessment tool during the study

SUMMARY:
This is a prospective descriptive monocentric study whose purpose is to describe the clonal evolution of the mutational pattern in cfDNA of a cohort of patients with Diffuse Large B-Cell Non-Hodgkin Lymphomas (DLBCL) before, during and after standard treatment

DETAILED DESCRIPTION:
To determinate and to describe the clonal evolution, 30 DLBCL cases with available matched tumor DNA and plasma will be collected and analyzed by routinely applicable next generation sequencing (NGS) at the time of diagnosis, at mid treatment, at the end of treatment and at 12 months after diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age up to 18 years old
* With a diagnosis formally established of DLBCL or transformed straightaway follicular lymphoma or 3B grade follicular lymphoma or Burkitt-like lymphoma
* Eligible to a treatment by immunochemotherapy like R-CHOP, R-ACVBP or R-CHOP like
* First line of treatment
* Being able to benefit from standard extension assessment ( Fluorine-18 fluorodeoxyglucose positron emission tomography (18F-FDG-PET) and bone marrow biopsy with a bone marrow aspiration)
* Written informed consent
* Tumor biopsy used for diagnosis available

Exclusion Criteria:

* Patient who cannot receive polychemotherapy like R-CHOP, R-ACVBP, or R-CHOP like
* Patient who cannot benefit from standard extension assessment and follow-up by with Fluorine-18 fluorodeoxyglucose positron emission tomography (18F-FDG-PET)
* Pregnant or breast-feeding woman
* Guardianship, curatorship
* Patient who cannot follow the medical procedures of the study for geographic, social, psychological,linguistic or physical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Determine the clonal evolution during and after treatment by Next Generation Sequencing | one year
  DNA from tumor, DNA from peripheral blood and DNA from bone marrow will be sequencing by NGS for a panel of 34 genes.

SECONDARY OUTCOMES:
Progression free survival | One year
  time between inclusion and progression or relapse or beginning of a new treatment
Overall survival | one year
  time between inclusion and death
Assess the clonal architecture in tumor DNA and bone marrow | one year
Compare the Fluorine-18 fluorodeoxyglucose positron emission tomography (18F-FDG-PET) procedure and the kinetic and pattern of somatic mutations identified in cfDNA | one year

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Jardin, Professor, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

REFERENCES:
- [Derived] Camus V, Sarafan-Vasseur N, Bohers E, Dubois S, Mareschal S, Bertrand P, Viailly PJ, Ruminy P, Maingonnat C, Lemasle E, Stamatoullas A, Picquenot JM, Cornic M, Beaussire L, Bastard C, Frebourg T, Tilly H, Jardin F. Digital PCR for quantification of recurrent and potentially actionable somatic mutations in circulating free DNA from patients with diffuse large B-cell lymphoma. Leuk Lymphoma. 2016 Sep;57(9):2171-9. doi: 10.3109/10428194.2016.1139703. Epub 2016 Feb 17. PMID 26883583